CLINICAL TRIAL: NCT07271420
Title: Blood Pressure Control With Thiazide Diuretics in Peritoneal Dialysis Patients
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Chan Chun Kau Gordon, Dr, Chinese University of Hong Kong
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CREC2019.580
Record Dates: First submitted 2025-11-26; First posted 2025-12-09 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-11

CONDITIONS: Hypertension; Peritoneal Dialysis; End Stage Kidney Disease (ESRD)
Keywords: Hypertension; Thiazides diuretics; End stage kidney disease; Peritoneal dialysis
MeSH Terms: conditions — Hypertension; Kidney Failure, Chronic | interventions — Hydrochlorothiazide

STUDY DESIGN:
Intervention Model Description: Following written informed consent, participants entered the treatment arm, receiving oral hydrochlorothiazide once daily on top of their standard of treatment for 90 days. This was followed by a 14-day washout period, after which participants entered a 90-day control period.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Thiazides treatment arm (Active Comparator)
  Interventions: Drug: Hydrochlorothiazide 25mg once per day
- Control arm (No Intervention)

INTERVENTIONS:
Drug: Hydrochlorothiazide 25mg once per day — Thiazides diuretics
  Arms: Thiazides treatment arm

SUMMARY:
To evaluate the blood pressure lowering effects of thiazide diuretics in patients on peritoneal dialysis

DETAILED DESCRIPTION:
This prospective, single-center treatment-withdrawal crossover study enrolled 10 patients on chronic peritoneal dialysis (PD) and uncontrolled hypertension (SBP >140 mmHg and/or DBP >90 mmHg).

Following written informed consent, participants entered the treatment arm, receiving oral hydrochlorothiazide once daily on top of their standard of treatment for 90 days. This was followed by a 14-day washout period, after which participants entered a 90-day control period.

ELIGIBILITY:
Inclusion Criteria:

* Patients on chronic peritoneal dialysis, with uncontrolled hypertension (SBP >140 mmHg and/or DBP >90 mmHg)

Exclusion Criteria:

* Patients with a life expectancy of less than 3 months, planned conversion to hemodialysis, or scheduled kidney transplantation within 3 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2020-01-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Change in systolic and diastolic blood pressure | 90 days

SECONDARY OUTCOMES:
Changes in body weight | 90 days
Changes in body composition measured by bio impedance spectroscopy | 90 days
Change in urinary fractional excretion of sodium | 90 days

CONTACTS AND LOCATIONS:
Locations (1):
- Prince of Wales Hospital. The Chinese University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No
Additional consent will need to be obtained from the participants

REFERENCES:
- [Background] Agarwal R, Sinha AD, Cramer AE, Balmes-Fenwick M, Dickinson JH, Ouyang F, Tu W. Chlorthalidone for Hypertension in Advanced Chronic Kidney Disease. N Engl J Med. 2021 Dec 30;385(27):2507-2519. doi: 10.1056/NEJMoa2110730. Epub 2021 Nov 5. PMID 34739197
- [Background] Ali S, Navaneethan SD, Virani SS, Gregg LP. Revisiting diuretic choice in chronic kidney disease. Curr Opin Nephrol Hypertens. 2022 Sep 1;31(5):406-413. doi: 10.1097/MNH.0000000000000814. Epub 2022 Jul 11. PMID 35894274
- [Background] An J, Kurella Tamura M, Odden MC, Ni L, Thomas IC, Montez-Rath ME, Sim JJ. Prevalence of Apparent Treatment-Resistant Hypertension in Chronic Kidney Disease in Two Large US Health Care Systems. Clin J Am Soc Nephrol. 2022 Oct;17(10):1457-1466. doi: 10.2215/CJN.04110422. Epub 2022 Sep 9. PMID 36400564
- [Background] Chan GC, Ng JK, Chow KM, Cheng PM, Law MC, Leung CB, Li PK, Szeto CC. Polypharmacy Predicts Onset and Transition of Frailty, Malnutrition, and Adverse Outcomes in Peritoneal Dialysis Patient. J Nutr Health Aging. 2022;26(12):1054-1060. doi: 10.1007/s12603-022-1859-8. PMID 36519768